CLINICAL TRIAL: NCT03427580
Title: Metacognitive and Insight Therapy (MERIT) for Persons With Schizophrenia: Assessment of Session by Session Progress and Outcome.
Brief Title: Metacognitive and Insight Therapy for Persons With Schizophrenia (RCT MERIT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bar-Ilan University, Israel (Other)
Responsible Party: Principal Investigator, Ilanit Hasson-Ohayon, Prof. Ilanit Hasson-Ohayon, Principal Investigator, Bar-Ilan University, Israel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MERIT
Record Dates: First submitted 2018-02-04; First posted 2018-02-09 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Diagnosis of Schizophrenia Spectrum Disorders
Keywords: Schizophrenia; Psychotherapy; Metacognitive abilities; Session by session assessment; Outcome
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental)
  Interventions: Behavioral: MERIT
- delayed treatment control group (Experimental)
  Interventions: Behavioral: MERIT

INTERVENTIONS:
Behavioral: MERIT — Metacognitive Reflection and Insight Therapy

SUMMARY:
People with schizophrenia spectrum disorders are faced with significant metacognitive impairments that include difficulties in their ability to form complex representations of the self and others. These impairments are associated with increased symptoms, impaired subjective self-experiences, and lower social functioning. As a result, interventions that enhance metacognitive capacity have been recently developed and explored. One of these interventions is Metacognitive Reflection and Insight Therapy (MERIT; Lysaker et al., 2014). MERIT is an integrative model of psychotherapy that seeks to promote holistic metacognitive capacity and consequently increase a positive sense of agency and sense of meaning in life among clients with schizophrenia. Several case studies (including in Bar-Ilan's community clinic), as well as a recent pilot study, showed increased metacognitive abilities and a decrease in symptoms following MERIT. The current study will explore both the effectiveness and the change mechanisms that underlie MERIT interventon among clients diagnosed with schizophrenia spectrum disorders, via both pre- and post-measures of the intervention's outcome and session-by-session estimations of the therapeutic process.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia spectrum disorders
* Ability to provide informed consent
* Ability to read and write in Hebrew

Exclusion Criteria:

* No co-morbid nuerological condition
* No hospitalization in the last 6 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bar-Ilan University, Ramat Gan, Israel

REFERENCES:
- [Derived] Lavi-Rotenberg A, Bar-Kalifa E, de Jong S, Igra L, Lysaker PH, Hasson-Ohayon I. Elements that enhance therapeutic alliance and short-term outcomes in metacognitive reflection and insight therapy: A session-by-session assessment. Psychiatr Rehabil J. 2020 Dec;43(4):318-326. doi: 10.1037/prj0000415. Epub 2020 Apr 9. PMID 32271073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were 35 adults diagnosed with of schizophrenia /schizoaffective disorder. Exclusion criteria: intellectual disability, neurological disorders, substance use problems, acute psychosis, and risk for suicidal behavior, based on the intake interview.
  The study used a delayed randomized controlled trial design to examine the therapeutic benefits of MERIT delivered in a community clinic at Bar-Ilan University.
Period: Overall Study
Arm/Group | Treatment Group | Delayed Treatment Control Group
Started | 31 | 23
Completed | 21 | 14
Not Completed | 10 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Delayed Treatment Control Group | Total
Number analyzed (Participants) | 31 | 23 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (10.63) | 40.5 (8.71) | 39.6 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 13 | 9 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: The number analyzed in row differs from overall due to dropouts.
  participants
    Israel: number analyzed (Participants) | 21 | 14 | 35
    Israel | 21 | 14 | 35

OUTCOME MEASURES:

1. Primary Outcome: Metacognition Assessment Scale-Abbreviated (MAS-A)
Description: The Metacognition Assessment Scale-Abbreviated (MAS-A) is a rating scale used to assess metacognitive abilities in individuals, particularly those with psychiatric conditions. The scale consists of four domains that reflect one's ability to understand different mental phenomena and use this understanding in order to cope with psychological challenges.
  Higher scores indicate a higher complexity of functions and ideas in each domain, i.e. higher values represent a better outcome. The four scales/domains:
  1. self-reflectivity (min 1 to max 9) ;
  2. understanding of the other's mind (min 1 to max 7) ;
  3. decentration (min 1 to max 3) ;
  4. mastery (min 1 to max 9). The total score is the sum of the ratings in each subscale. Thus, the total score can be ranged from 4 (min) to 28 (max), when higher values represent a better outcome.
Time Frame: Prior to the begining of the therapy (baseline, pre-treatment), and again at the end of the therapy (six months later, post-treatment)
Population: The N in the "POST" row is following dropouts.
  Treatment Group Arm: Baseline/pre-treatment and post-treatment at 24 weeks; For Delayed Treatment Control Group Arm: Baseline/pre-waiting period and 6 months post-waiting period prior to starting treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delayed Treatment Control Group | Treatment Group
Number analyzed (Participants) | 31 | 23
score on a scale
  Pre (treatment/waiting period) | 11.53 (3.7) | 14.22 (2.75)
  Post (treatment/waiting period): number analyzed (Participants) | 21 | 14
  Post (treatment/waiting period) | 14.22 (3.4) | 14.25 (4.2)

ADVERSE EVENTS:
Time Frame: 2 years
Description: The definition of adverse event and/or serious adverse event does not differ from the clinicaltrials.gov Definitions.
Arm/Group | Treatment Group | Delayed Treatment Control Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/23
Other Adverse Events (participants affected / at risk) | 0/31 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT03427580/Prot_SAP_000.pdf